CLINICAL TRIAL: NCT05751421
Title: Comparing the Efficacy of a Periarticular Instillation of Extended Relief Bupivacaine and Meloxicam With Routine Adductor Canal Blockade for Pain Relief After Primary TKA
Brief Title: Pain Relief After PrimaryTKA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iRIS1128_JLON
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — bupivacaine-meloxicam drug combination; Bupivacaine; Meloxicam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- primary total knee replacement + Zynrelef (Experimental): Patients undergoing primary total knee replacement with Extended Relief Bupivacaine and Meloxicam (Zynrelef)
  Interventions: Drug: Zynrelef (Bupivacaine 60 MG / Meloxicam 1.8 MG) Per 2.3 ML Extended Release Solution; Procedure: primary total knee replacement
- primary total knee replacement + adductor canal block (ACB) (Active Comparator): Patients undergoing primary total knee replacement with routine adductor canal block
  Interventions: Drug: Bupivacaine HCl 0.5% Injectable Solution; Procedure: primary total knee replacement

INTERVENTIONS:
Drug: Zynrelef (Bupivacaine 60 MG / Meloxicam 1.8 MG) Per 2.3 ML Extended Release Solution — zynrelef will be administered during surgery
  Arms: primary total knee replacement + Zynrelef
Drug: Bupivacaine HCl 0.5% Injectable Solution — adductor canal block will be performed using bupivacaine before surgery
  Arms: primary total knee replacement + adductor canal block (ACB)
Procedure: primary total knee replacement — primary total knee replacement

SUMMARY:
While a majority of people who undergo TKA have significant long-term improvement in functional ability, many patients may experience significant pain in the early postoperative period, which may adversely impact postoperative rehabilitation and recovery. Traditionally, opioid medications have been used to control postoperative pain. However, there are many risks with using opioid medications, including addiction and overdose, which kills over 48,000 people yearly. In an effort to overcome this, opioid-sparing multimodal analgesia (MMA) regimens have been developed, commonly using nonsteroid anti-inflammatory drugs (NSAIDs), acetaminophen, regional nerve blocks, and local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Patients undergoing primary unilateral TKA
* Patients receiving spinal anesthesia during primary TKA
* Patients with adequate cognitive function to participate and complete questionnaires for the study

Exclusion Criteria:

* Patients undergoing bilateral simultaneous TKA
* Patients undergoing conversion TKA
* Patients undergoing unicompartmental knee arthroplasty
* Patients undergoing patellofemoral arthroplasty
* Patients with an allergy to NSAIDs or bupivacaine
* Patients who have a contraindication to the use of NSAIDs
* Patients who are using chronic anticoagulation, precluding them from using NSAIDs
* Patients with a history or diagnosis of chronic pain syndrome or complex regional pain syndrome
* Patients who are determined to be in severe pain from other concomitant conditions
* Patients with chronic opioid use disorder, defined as patients who are taking more than 20 mg/day morphine milligram equivalents for 30 days consecutively in the 3 months prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 14 days
  This will be measured by a postoperative Visual Analog Score (VAS) completed by the participant
Opioid consumption | 14 days
  Participants will be asked to keep a diary of how much pain medication they took after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States